CLINICAL TRIAL: NCT06085859
Title: Anesthesia Endoscope Mask is Applied to Sedation Upper Gastrointestinal Endoscopic Diagnosis and Treatment: Multi-center, Prospective, Randomized Control, Open Clinical Research
Brief Title: Anesthesia Endoscope Mask is Applied to Sedation Upper Gastrointestinal Endoscopic Diagnosis and Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Collaborators: Anhui Sanhong Medical Device Technology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Mengchang Yang, Principal Investigator, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: endoscope mask-1
Record Dates: First submitted 2023-09-25; First posted 2023-10-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hypoxemia
Keywords: hypoxemia; sedation; gastrointestinal sedation procedure; non-invasive ventilation; endoscopy mask
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Randomly assign participants to the standard nasal catheter oxygenation group and the endoscopy mask oxygen inhalation group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mask oxygen supply group (Experimental): The anaesthesia provider supplied oxygen via a nasal cannula at an oxygen flow rate of 8 Litres/minute supplied from an oxygen flowmeter
  Interventions: Device: Mask group
- Nasal oxygen supply group (Experimental): The study team applied the mask with a head strap to ensure a proper seal,simultaneously ensuring the same oxygen flow rate as the control group
  Interventions: Device: Routine nasal catheter group

INTERVENTIONS:
Device: Routine nasal catheter group — The anaesthesia provider supplied oxygen via a nasal cannula at an oxygen flow rate of 8 Litres/minute supplied from an oxygen flowmeter as described in the guide
  Arms: Nasal oxygen supply group
Device: Mask group — The study team applied the mask with a head strap to ensure a proper seal,simultaneously ensuring the same oxygen flow rate as the control group
  Arms: Mask oxygen supply group

SUMMARY:
To investigate the efficacy and safety of new-type mask compared with nasal tube oxygen delivery in patients undergoing sedation of upper gastrointestinal endoscopy

DETAILED DESCRIPTION:
This study aims to utilize a large sample, multicenter, prospective clinical trial using a new mask oxygen supply technology. If the study confirms that the new mask can improve the airway safety and effectiveness in patient examinations, while improving examination efficiency and reducing failure rates, it will provide safety assurance for the early diagnosis and treatment of upper gastrointestinal diseases in high-risk populations.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Upcoming upper gastrointestinal sedation procedure;
3. Classification under the American Association of Anesthesiologists (ASA) status I-III;
4. Baseline oxygen saturation (SpO2) ≥95% in ambient air conditions.

Exclusion Criteria:

1. Individuals with previously documented difficulties in mask ventilation (DMV);
2. Patients predisposed to aspiration risks or episodes of vomiting;
3. Facial or jaw injuries or congenital abnormalities that render conventional face mask application infeasible;
4. An inability or unwillingness to utilize the novel disposable anesthesia face mask.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1208 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypoxemia | From the start of drug administration by the researcher to the completely withdraw from the endoscopy by the end of the examination.
  Incidences of oxygen saturation falling below 92%

SECONDARY OUTCOMES:
Incidence of compromised ventilation mandating primary manual intervention | From the start of drug administration by the researcher to the completely withdraw from the endoscopy by the end of the examination.
  For the nasal catheter cohort, this entailed jaw elevation and deploying a standard mask to augment the oxygen concentration inhaled. Concurrently, for the mask cohort, primary intervention involved mandible lifting and secure fastening of the mask sleeve for inflation (while ensuring the operational aperture remains sealed).
Incidence necessitating sophisticated manual ventilatory support during pain-free gastroscopy | From the start of drug administration by the researcher to the completely withdraw from the endoscopy by the end of the examination.
  If SpO2 levels further descended to ≤70% or persistently hovered below 85% for a duration exceeding 60 seconds, it mandated an immediate cessation of the ongoing procedure. The endoscope would be retracted, followed by the insertion of a standard oropharyngeal mask for assisted ventilation. In dire circumstances, the anesthesiologist might opt for advanced airway interventions, such as laryngeal mask application or endotracheal intubation.
Juxtaposition of hypoxemia onset time in both ventilation techniques | From the start of drug administration by the researcher to the completely withdraw from the endoscopy by the end of the examination.
  The time span from the start of drug administration by the researcher to the first occurrence of blood oxygen saturation below 92%.
the temporal span from initial decline to recovery to 92% saturation in both ventilation techniques | From the start of drug administration by the researcher to the completely withdraw from the endoscopy by the end of the examination.
  The time span from oxygen saturation below 92% to recovery to 92% after manual ventilatory support. If multiple episodes of hypoxia occur, all times will be added up
the lowest oxygen saturation in both ventilation techniques | From the start of drug administration by the researcher to the completely withdraw from the endoscopy by the end of the examination.
  the lowest oxygen saturation from the start of medication administration to the participants's Aldrete score of 9.
Evaluation of procedural prolongation due to ventilation issues | From the start of drug administration by the researcher to the completely withdraw from the endoscopy by the end of the examination.
  The extension time for examination is defined as the total time from stopping the operation and exiting the endoscope until the endoscope re-enters the digestive tract, to the same anatomical position before stopping the operation, If multiple episodes of withdrawal of endoscopy occur, all times will be added up
Apnea prevalence in both groups | From the start of drug administration by the researcher to the completely withdraw from the endoscopy by the end of the examination.
  The study here we define apnea as 10 second without obvious respiratory movements of mesothorax and abdomen or snoring with paradoxical breathing
Satisfaction scores1 from patients, endoscopists, and anesthesiologists | Immediately after the procedure.
  The scores of satisfaction 1：Are you satisfied with this endoscopic diagnosis and treatment,a score of 0 represents very dissatisfied, while a score of 10 represents very satisfied.
Satisfaction scores2 from patients, endoscopists, and anesthesiologists | Immediately after the procedure.
  The scores of satisfaction2：If there is a chance, are you willing to use this non-invasive oxygen device again,a score of 0 indicates a strong unwillingness, while a score of 10 indicates a strong willingness.
The incidence of upper respiratory tract discomfort manifestations such as oral, nasal, an pharyngeal dryness and hemorrhage in two groups of participants. | Immediately after the procedure.
Inaugural insertion success rates in two groups of participants | From the start of drug administration by the researcher to the completely withdraw from the endoscopy by the end of the examination.
  If the endoscopic operation fails to pass the pharynx after three attempts, recorded as the first insertion failure.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - First People's Hospital of Liangshan Yi Autonomous Prefecture, Liangshan, Sichuan
  - Second People's Hospital of Yibin, Yibin, Sichuan
  - Ziyang People's Hospital, Ziyang, Sichuan
  - Chengdu Second People's Hospital, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
After December 2024, the original data can be obtained through the author's email address.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After December 2024
Access Criteria: Any project applicant

REFERENCES:
- [Background] Behrens A, Kreuzmayr A, Manner H, Koop H, Lorenz A, Schaefer C, Plauth M, Jetschmann JU, von Tirpitz C, Ewald M, Sackmann M, Renner W, Kruger M, Schwab D, Hoffmann W, Engelke O, Pech O, Kullmann F, Pampuch S, Lenfers B, Weickert U, Schilling D, Boehm S, Beckebaum S, Cicinnati V, Erckenbrecht JF, Dumoulin FL, Benz C, Rabenstein T, Haltern G, Balsliemke M, de Mas C, Kleber G, Pehl C, Vogt C, Kiesslich R, Fischbach W, Koop I, Kuehne J, Breidert M, Sass NL, May A, Friedrich C, Veitt R, Porschen R, Ellrichmann M, Arlt A, Schmitt W, Dollhopf M, Schmidbaur W, Dignass A, Schmitz V, Labenz J, Kaiser G, Krannich A, Barteska N, Ell C. Acute sedation-associated complications in GI endoscopy (ProSed 2 Study): results from the prospective multicentre electronic registry of sedation-associated complications. Gut. 2019 Mar;68(3):445-452. doi: 10.1136/gutjnl-2015-311037. Epub 2018 Jan 3. PMID 29298872
- [Background] Nay MA, Fromont L, Eugene A, Marcueyz JL, Mfam WS, Baert O, Remerand F, Ravry C, Auvet A, Boulain T. High-flow nasal oxygenation or standard oxygenation for gastrointestinal endoscopy with sedation in patients at risk of hypoxaemia: a multicentre randomised controlled trial (ODEPHI trial). Br J Anaesth. 2021 Jul;127(1):133-142. doi: 10.1016/j.bja.2021.03.020. Epub 2021 Apr 28. PMID 33933271
- [Background] Goudra B, Nuzat A, Singh PM, Borle A, Carlin A, Gouda G. Association between Type of Sedation and the Adverse Events Associated with Gastrointestinal Endoscopy: An Analysis of 5 Years' Data from a Tertiary Center in the USA. Clin Endosc. 2017 Mar;50(2):161-169. doi: 10.5946/ce.2016.019. Epub 2016 Apr 29. PMID 27126387
- [Background] Qin Y, Li LZ, Zhang XQ, Wei Y, Wang YL, Wei HF, Wang XR, Yu WF, Su DS. Supraglottic jet oxygenation and ventilation enhances oxygenation during upper gastrointestinal endoscopy in patients sedated with propofol: a randomized multicentre clinical trial. Br J Anaesth. 2017 Jul 1;119(1):158-166. doi: 10.1093/bja/aex091. PMID 28974061
- [Background] Bell GD, Bown S, Morden A, Coady T, Logan RF. Prevention of hypoxaemia during upper-gastrointestinal endoscopy by means of oxygen via nasal cannulae. Lancet. 1987 May 2;1(8540):1022-4. doi: 10.1016/s0140-6736(87)92282-3. PMID 2883355
- [Background] Terblanche NCS, Middleton C, Choi-Lundberg DL, Skinner M. Efficacy of a new dual channel laryngeal mask airway, the LMA(R)Gastro Airway, for upper gastrointestinal endoscopy: a prospective observational study. Br J Anaesth. 2018 Feb;120(2):353-360. doi: 10.1016/j.bja.2017.11.075. Epub 2017 Dec 1. PMID 29406183
- [Background] King AB, Alvis BD, Hester D, Taylor S, Higgins M. Randomized trial of a novel double lumen nasopharyngeal catheter versus traditional nasal cannula during total intravenous anesthesia for gastrointestinal procedures. J Clin Anesth. 2017 May;38:52-56. doi: 10.1016/j.jclinane.2017.01.025. Epub 2017 Jan 22. PMID 28372678
- [Background] Hung KC, Chang YJ, Chen IW, Soong TC, Ho CN, Hsing CH, Chu CC, Chen JY, Sun CK. Efficacy of high flow nasal oxygenation against hypoxemia in sedated patients receiving gastrointestinal endoscopic procedures: A systematic review and meta-analysis. J Clin Anesth. 2022 May;77:110651. doi: 10.1016/j.jclinane.2022.110651. Epub 2022 Jan 12. PMID 35030538